CLINICAL TRIAL: NCT02194283
Title: A Double-blind (at Each Dose Level), Randomised, Placebo Controlled Phase I Study to Evaluate Safety, Tolerability and Pharmacokinetics of Increasing Repeated Oral Doses of Ambroxol Lozenges (Dosage: 20, 40, 80 mg Three Times Daily) Over 4 Days in Healthy Male Volunteers
Brief Title: Study to Evaluate Safety, Tolerability and Pharmacokinetics of Increasing Repeated Oral Doses of Ambroxol Lozenges in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 18.493
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Ambroxol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ambroxol - in single rising doses (Experimental)
  Interventions: Drug: Ambroxol - in single rising doses
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ambroxol - in single rising doses
  Arms: Ambroxol - in single rising doses
Drug: Placebo
  Arms: Placebo

SUMMARY:
The main objectives of the present study are to determine pharmacokinetics of ambroxol in healthy male volunteers following repeated administration of lozenges of 20 mg ambroxol for four days

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs, 12-lead Electrocardiogram (ECG), clinical laboratory tests
* Age ≥21 and Age ≤50 year
* BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including vital signs and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Actual smoker
* Alcohol abuse (more than 40 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalaemia, family history of Long QT Syndrome)

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 24 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 24 hours after drug administration
AUC0-24 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 hours) | up to 24 hours after drug administration
Ae0-24 (amount of the analyte that is eliminated in urine from the time point 0 until time point 24) | up to 24 hours after drug administration
CLR,0-24 (renal clearance of the analyte determined from the time point 0 until time point 24) using AUC0-24 and Ae0-24 | up to 24 hours after drug administration
Cmax,ss (maximum concentration of the analyte in plasma at steady state) | up to 120 hours after first drug administration
tmax,ss (time from last dosing to maximum concentration at steady state) | up to 120 hours after first drug administration
Cmin,ss (minimum concentration of the analyte in plasma at steady state) | up to 120 hours after first drug administration
AUC72-96,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform 24 hour interval matching Day 1) | up to 96 hours after first drug administration
Ae72-96,ss (amount of analyte that is eliminated in urine at steady state from the time point 72 to time point 96) | up to 96 hours after first drug administration
CLR,72-96,ss (renal clearance of the analyte in plasma from the time point 72 until the time point 96 at steady state) using AUC72-96 and Ae72-96 | up to 96 hours after first drug administration
λz,ss (terminal rate constant in plasma at steady state) | up to 120 hours after first drug administration
t1/2,ss (terminal half-life of the analyte in plasma at steady state) | up to 120 hours after first drug administration
RA (accumulation ratio) | up to 96 hours after first drug administration
LI (linearity index) | up to 96 hours after first drug administration

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 36 days
Number of patients with abnormal changes in laboratory parameters | up to 36 days
Number of patients with clinically significant changes in vital signs (blood pressure [BP], pulse rate [PR]) | up to 36 days
Number of patients with clinically significant changes in 12-lead electrocardiogram (ECG) | up to 36 days
Assessment of tolerability on a 4-point scale | 10 days after last drug administration